CLINICAL TRIAL: NCT04026113
Title: A Phase 3, Multicenter, Randomized, Double-blind, Parallel-group, Safety and Efficacy Study of Linaclotide in Pediatric Participants, Ages 6 to 17 Years, With Irritable Bowel Syndrome With Constipation (IBS-C) and of Linaclotide Versus Placebo in Pediatric Participants With Functional Constipation (FC)
Brief Title: Linaclotide Safety and Efficacy in Pediatric Participants, 6 to 17 Years of Age, With Irritable Bowel Syndrome With Constipation (IBS-C) or Functional Constipation (FC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIN-MD-64; 2019-001500-38 (EudraCT Number)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Functional Constipation; Irritable Bowel Syndrome With Constipation
Keywords: Functional constipation in children; Irritable Bowel Syndrome with Constipation; LINZESS
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- FC Participants: Placebo (Experimental): Placebo single dose, once daily at approximately the same time each day, 30 minutes before any meal.
  Interventions: Drug: Placebo
- FC Participants: Linaclotide 72 μg (Experimental): Linaclotide 72 μg single dose, once daily at approximately the same time each day, 30 minutes before any meal.
  Interventions: Drug: Linaclotide
- IBS-C Participants: Linaclotide 145 μg (Experimental): Linaclotide 145 μg single dose, once daily at approximately the same time each day, 30 minutes before any meal.
  Interventions: Drug: Linaclotide
- IBS-C Participants: Linaclotide 290 μg (Experimental): Linaclotide 290 μg single dose, once daily at approximately the same time each day, 30 minutes before any meal
  Interventions: Drug: Linaclotide

INTERVENTIONS:
Drug: Linaclotide — Oral capsule (For participants who do not wish to take the dose as a capsule, a sprinkled dose may be prepared)
  Arms: FC Participants: Linaclotide 72 μg; IBS-C Participants: Linaclotide 145 μg; IBS-C Participants: Linaclotide 290 μg
Drug: Placebo — Matching placebo
  Arms: FC Participants: Placebo

SUMMARY:
The objective of LIN-MD-64 is to evaluate the safety and efficacy of 12 weeks of linaclotide therapy (72 μg daily) in comparison with placebo in pediatric participants, 6 to 17 years of age, who fulfill modified Rome III Criteria for child/adolescent FC. The objective of LIN-MD-64 is to evaluate the safety and efficacy of 12 weeks of linaclotide therapy (145 μg or 290 μg daily) in pediatric participants 7 to 17 years of age, who fulfill the Rome III criteria for child/adolescent IBS and modified Rome III criteria for child/adolescent FC.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be ages 6 to 17 years (FC participants) or ages 7 to 17 years (IBS-C participants) (inclusive) at the time the participant provides assent for the study and parent/guardian/legally authorized representative (LAR) has provided signed consent;
* Participant weighs ≥18 kg at the time the participant provides assent and the parent/guardian/LAR has provided signed consent;
* Participants who meet the modified Rome III criteria for Child/Adolescent FC. For at least 2 months before the Screening Visit, the participant has had 2 or fewer defecations (with each defecation occurring in the absence of any laxative, suppository, or enema use during the preceding 24 hours) in the toilet per week.

In addition, participant meets one or more of the following criteria at least once per week for at least 2 months before the screening visit:

a. History of retentive posturing or excessive volitional stool retention; b. History of painful or hard BMs; c. History of large diameter stools that may obstruct the toilet; d. Presence of a large fecal mass in the rectum; e. At least 1 episode of fecal incontinence per week

* For IBS-C participants only: Participant meets Rome III criteria for child/adolescent IBS: At least once per week for at least 2 months before the Screening Visit, the participant experienced abdominal discomfort (an uncomfortable sensation not described as pain) or pain associated with 2 or more of the following at least 25% of the time:

  1. Improvement with defecation;
  2. Onset associated with a change in frequency of stool;
  3. Onset associated with a change in form (appearance) of stool;
* For IBS-C participants only: Participant has an average daytime abdominal pain score of ≥ 1 (at least "a tiny bit") during the 14 days before Visit 3;
* Participant is willing to discontinue any laxatives used before the Preintervention Visit in favor of the protocol- permitted rescue medicine;
* Participant has an average of fewer than 3 SBMs per week during the 14 days before the randomization day and up to the randomization (including the morning eDiary assessments reported before administration of first dose of double-blind study intervention on the randomization day). An SBM is defined as a BM that occurs in the absence of laxative, enema, or suppository use on the calendar day of the BM or the calendar day before the BM;
* Participant or parent/guardian/LAR or caregiver is compliant with eDiary requirements by completing both the morning and evening assessments for 10 out of the 14 days immediately preceding the Randomization Visit;
* Female participants of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Randomization Visit prior to dosing;
* Female participants who have had their first menstrual period and are sexually active must agree to use a reliable form of contraception;
* Participant must provide written or verbal informed assent and the parent/guardian/LAR and caregiver must provide written informed consent before the initiation of any study-specific procedures;
* Participant is able to read and/or understand the assessments in the eDiary device. If the participant is 6 to 11 years of age (FC participants) or 7 to 11 years of age (IBS-C participants) and does not meet this criterion, the interviewer-administered version of the eDiary must be used and the parent/guardian/LAR or caregiver who will be administering the interviewer-administered version of the eDiary must undergo training;
* Participant must have acquired toilet training skills.

Exclusion Criteria:

* For FC participants only: Participant meets Rome III criteria for Child/Adolescent IBS: At least once per week for at least 2 months before the Screening Visit, the participant has experienced abdominal discomfort (an uncomfortable sensation not described as pain) or pain associated with 2 or more of the following at least 25% of the time:

  1. Improvement with defecation
  2. Onset associated with a change in frequency of stool
  3. Onset associated with a change in form (appearance) of stool;
* Participant reports having more than 1 loose, mushy stool (eDiary-recorded stool consistency of 6 on the Pediatric Bristol Stool Form Scale [p-BSFS]) or any watery stool (eDiary-recorded stool consistency of 7 on the p-BSFS) with any SBM that occurred in the absence of laxative use on the calendar day of the BM or the calendar day before the BM during the 14 days before the randomization day and up to the randomization (including the morning eDiary assessments reported before administration of first dose of double-blind study intervention on the randomization day);
* Participant has a history of non-retentive fecal incontinence;
* Participant has (a) fecal impaction at Visit 2 after failing outpatient clean-out during the Screening Period or (b) fecal impaction at Visit 3;
* Participant has required manual disimpaction any time prior to randomization;
* Participant currently has both unexplained and clinically significant alarm symptoms (lower GI bleeding [rectal bleeding or heme-positive stool], iron-deficiency anemia, or any unexplained anemia, or weight loss) and systemic signs of infection or colitis, or any neoplastic process;
* Participant has clinically significant findings on a physical examination, vital sign assessment, electrocardiogram (ECG), or clinical laboratory test as determined by the investigator based on consideration of whether the finding could represent a safety concern or a condition that would be exclusionary, could prevent the participant from performing any protocol assessments, or could confound study assessments;
* Participant has a history of drug or alcohol abuse;
* Participant has any of the following conditions:

  1. Celiac disease, or positive serological test for celiac disease and the condition has not been ruled out by endoscopic biopsy;
  2. Cystic fibrosis;
  3. Hypothyroidism that is untreated or treated with thyroid hormone at a dose that has not been stable for at least 3 months prior to the Screening Visit;
  4. Down's syndrome or any other chromosomal disorder;
  5. Active anal fissure (Note: History of anal fissure is not an exclusion);
  6. Anatomic malformations (eg, imperforate anus, anal stenosis, anterior displaced anus);
  7. Intestinal nerve or muscle disorders (eg, Hirschprung disease, visceral myopathies, visceral neuropathies);
  8. Neuropathic conditions (eg, spinal cord abnormalities, neurofibromatosis, tethered cord, spinal cord trauma);
  9. Lead toxicity, hypercalcemia;
  10. Neurodevelopmental disabilities (early-onset, chronic disorders that share the essential feature of a predominant disturbance in the acquisition of cognitive, motor, language, or social skills, which has a significant and continuing impact on the developmental progress of an individual) producing a cognitive delay that precludes comprehension and completion of the daily eDiary (Electronic handheld device) or other study-related questionnaires (Note: Participants are excluded if the person who will be completing the daily eDiary or other study-related questionnaires meets this criterion);
  11. Inflammatory bowel disease;
  12. Childhood functional abdominal pain syndrome;
  13. Childhood functional abdominal pain;
  14. Poorly treated or poorly controlled psychiatric disorders that might influence his or her ability to participate in the study;
  15. Lactose intolerance that is associated with abdominal pain or discomfort and could confound the assessments in this study;
  16. History of cancer other than treated basal cell carcinoma of the skin; (Note: Participants with a history of cancer are allowed provided that the malignancy has been in a complete remission for at least 5 years before the Randomization Visit. A complete remission is defined as the disappearance of all signs of cancer in response to treatment);
  17. History of diabetic neuropathy.
* Participant has an acute or chronic condition that, in the investigator's opinion, would limit the participants' ability to complete or participate in this clinical study;
* Participant has a known or suspected mechanical bowel obstruction or pseudoobstruction;
* Participant has a known allergy or sensitivity to the study intervention or its components or other medications in the same drug class.
* Participant has had surgery that meets any of the following criteria:

  1. Bariatric surgery for treatment of obesity, or surgery to remove a segment of the GI tract at any time before the Screening Visit;
  2. Surgery of the abdomen, pelvis, or retroperitoneal structures during the 6 months before the Screening Visit;
  3. An appendectomy or cholecystectomy during the 60 days before the Screening Visit;
  4. Other major surgery during the 30 days before the Screening Visit;
* Participant used a protocol-specified prohibited medicine before the start of the Preintervention Period or failed to meet the stable-dose requirements of certain medications;
* Participant used rescue medication on the calendar day before the Randomization Visit and on the day of the Randomization Visit until randomized;
* Participant received a study intervention during the 30 days before the Screening Visit or is planning to receive a study intervention (other than that administered during this study);
* Participant has been randomized into any clinical study in which linaclotide was a study intervention.
* The participant has a condition or is in a situation; which, in the investigator's opinion, may put the participant at significant risk, may confound the study results ,or may interfere significantly with the participant's participation in the study;
* Participants who have positive urine drug screen results for cocaine, barbiturates, opiates, or cannabinoids will be excluded from study participation;
* Female participants who are currently pregnant or nursing, or plan to become pregnant or nurse during the clinical study;
* Participant's parent/guardian/LAR or caregiver has been directly or indirectly involved in the conduct and administration of this study as an investigator, study coordinator, or other study staff member. In addition, any participant, parent/guardian/LAR or caregiver who has a first-degree family member, significant other, or relative residing with him/her directly or indirectly who is involved in this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 438 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (115):
- United States (79):
  - Central Research Associates /ID# 233124, Birmingham, Alabama
  - G & L Research, LLC /ID# 233139, Foley, Alabama
  - The Center for Clinical Trials Inc. /ID# 232755, Saraland, Alabama
  - HealthStar Research of Hot Springs PLLC /ID# 232757, Hot Springs, Arkansas
  - Preferred Research Partners /ID# 233023, Little Rock, Arkansas
  - Applied Research Center of Arkansas /ID# 233135, Little Rock, Arkansas
  - Advanced Research Center /ID# 233121, Anaheim, California
  - Alliance Research Institute /ID# 232754, Bell Gardens, California
  - Alliance Research Institute Llc /Id# 232637, Canoga Park, California
  - Kindred Medical Institute, LLC /ID# 233042, Corona, California
  - Center for Clinical Trials LLC /ID# 232781, Paramount, California
  - Medical Ctr for Clin Research /ID# 233004, San Diego, California
  - Paragon Rx Clinical Inc /ID# 232752, Santa Ana, California
  - Lynn Institute of Denver /ID# 233137, Aurora, Colorado
  - Children's National Medical Center /ID# 232655, Washington D.C., District of Columbia
  - Prohealth Research Center /ID# 232805, Doral, Florida
  - Dolphin Medical Research /ID# 232815, Doral, Florida
  - Amedica Research Institute Inc /ID# 232809, Hialeah, Florida
  - Nemours Children's Health System /ID# 233127, Jacksonville, Florida
  - Elite Clinical Research /ID# 232801, Miami, Florida
  - My Preferred Research LLC /ID# 233119, Miami, Florida
  - South Miami Medical & Research Group Inc. /ID# 232803, Miami, Florida
  - Valencia Medical & Research Center /ID# 232813, Miami, Florida
  - Advanced Research for Health Improvement /ID# 233161, Naples, Florida
  - Pediatric & Adult Research Center /ID# 232819, Orlando, Florida
  - Nemours Children's Hospital /ID# 232919, Orlando, Florida
  - Oviedo Medical Research /ID# 232830, Oviedo, Florida
  - Treken Primary Care /ID# 232796, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Ferry Rd /ID# 233015, Atlanta, Georgia
  - Children's Ctr Digestive, US /ID# 233070, Atlanta, Georgia
  - River Birch Research Alliance /ID# 233122, Blue Ridge, Georgia
  - Clinical Research Institute /ID# 232833, Stockbridge, Georgia
  - Sleep Care Research Institute d/b/a Clinical Research Institute /ID# 232940, Stockbridge, Georgia
  - Clinical Trials Specialist Inc /ID# 232802, Stone Mountain, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG /ID# 232800, Union City, Georgia
  - Univ Kansas Med Ctr /ID# 232645, Kansas City, Kansas
  - Alliance for Multispecialty Research LLC /ID# 232681, Newton, Kansas
  - Michael W. Simon, MD, PSC /ID# 232966, Lexington, Kentucky
  - Meridian Research - Baton Rouge /ID# 232954, Baton Rouge, Louisiana
  - Virgo Carter Pediatrics /ID# 232693, Silver Spring, Maryland
  - MNGI Digestive Health, P. A. /ID# 232920, Minneapolis, Minnesota
  - GI associates and Endoscopy Ce /ID# 233123, Flowood, Mississippi
  - David M. Headley, MD, P.A. /ID# 233153, Port Gibson, Mississippi
  - Private Practice - Dr. Craig Spiegel /ID# 232707, Bridgeton, Missouri
  - Medclinical Research Partners LLC/ Foundation Pediatrics /ID# 232783, East Orange, New Jersey
  - University of New Mexico /ID# 233011, Albuquerque, New Mexico
  - Columbia Univ Medical Center /ID# 233094, New York, New York
  - The Children's Hospital at Montefiore /ID# 232638, The Bronx, New York
  - Advantage Clinical Trials /ID# 233117, The Bronx, New York
  - East Carolina University - Brody School of Medicine /ID# 233062, Greenville, North Carolina
  - PMG Research of Piedmont Healthcare-Statesville /ID# 233162, Statesville, North Carolina
  - Univ Oklahoma HSC /ID# 233067, Oklahoma City, Oklahoma
  - IPS Research Company /ID# 233081, Oklahoma City, Oklahoma
  - Frontier Clinical Research, LLC - Scottdale /ID# 233129, Scottdale, Pennsylvania
  - Frontier Clinical Research /ID# 233116, Smithfield, Pennsylvania
  - Rhode Island Hospital /ID# 233112, Providence, Rhode Island
  - Coastal Pediatric Research - West Ashley B /ID# 232816, Charleston, South Carolina
  - Coastal Pediatric Research - Summerville /ID# 232814, Summerville, South Carolina
  - The Jackson Clinic, PA /ID# 232998, Jackson, Tennessee
  - Accellacare of Knoxville /ID# 232663, Jefferson City, Tennessee
  - Monroe-Carell Jr. Children's Hospital at Vanderbilt /ID# 232659, Nashville, Tennessee
  - Oak Cliff Research Company LLC /ID# 232729, Dallas, Texas
  - Cook Children's Med. Center /ID# 233066, Fort Worth, Texas
  - Valley Institute of Research /ID# 232674, Harlingen, Texas
  - Vilo Research Group Inc /ID# 233155, Houston, Texas
  - Cullen Research /ID# 232726, Houston, Texas
  - Synergy Group US LLC /ID# 232669, Houston, Texas
  - Pioneer Research Solutions - Houston /ID# 233006, Houston, Texas
  - Synergy Group US LLC /ID# 232670, Missouri City, Texas
  - AIM Trials /ID# 232934, Plano, Texas
  - Sun Research Institute /ID# 233005, San Antonio, Texas
  - ClinPoint Trials /ID# 232978, Waxahachie, Texas
  - Chrysalis Clinical Research /ID# 232690, St. George, Utah
  - Office of Maria Ona /ID# 232700, Franklin, Virginia
  - Health Research of Hampton Roads, Inc. (HRHR) /ID# 233056, Newport News, Virginia
  - Clinical Research Partners, LLC /ID# 233026, Richmond, Virginia
  - Carilion Medical Center /ID# 232999, Roanoke, Virginia
  - Duplicate_Multicare Institute for Research and Innovation /ID# 233010, Tacoma, Washington
  - Marshall University Medical Center /ID# 232952, Huntington, West Virginia
- Duplicate_UZ Brussel /ID# 232875, Brussels, Belgium
- Bulgaria (4):
  - University Hospital Plovdiv /ID# 232775, Tsentar, Plovdiv
  - UMHAT Kanev /ID# 233102, Ruse, Smolyan
  - Medical center 1 Sevlievo /ID# 232915, Sevlievo, Smolyan
  - MHATSv.Ivan Rilski /ID# 232831, Kozloduy
- Canada (5):
  - University of Alberta Hospital /ID# 233147, Edmonton, Alberta
  - London Health Sciences Center- University Hospital /ID# 233068, London, Ontario
  - Duplicate_SKDS Research Inc. /ID# 233000, Newmarket, Ontario
  - Bluewater Clinical Research Group Inc /ID# 232772, Sarnia, Ontario
  - Stouffville Medical Centre /ID# 232774, Stouffville, Ontario
- Estonia (3):
  - Merelahe Family Doctors Centre /ID# 232881, Tallinn, Raplamaa
  - Kliiniliste Uuringute Keskus /ID# 232883, Tartu, Raplamaa
  - Al Mare Perearstikeskus /ID# 232879, Harjumaa
- Duplicate_Klinikum Kassel /ID# 233029, Kassel, Hesse, Germany
- Israel (7):
  - Schneider Children's Medical Center /ID# 233064, Petah Tikva, Central District
  - Duplicate_Rambam Health Care Campus Ruth Rappaport Children's Hospital /ID# 232892, Haifa, H_efa
  - Shaare Zedek Medical Center /ID# 233092, Jerusalem, Jerusalem
  - Hadassah Hebrew University Hospital - Ein Kerem /ID# 232865, Jerusalem, Jerusalem
  - The Baruch Padeh Medical Center Poriya /ID# 232889, Tiberias, Northern District
  - The Edith Wolfson Medical Center /ID# 233134, Ashkelon, Southern District
  - The Chaim Sheba Medical Center /ID# 232986, Ramat Gan, Tel Aviv
- Sant?Andrea University Hospital /ID# 232825, Rome, Italy
- Netherlands (3):
  - Duplicate_Academisch Medisch Centrum /ID# 232895, Amsterdam, North Holland
  - Maasstad Ziekenhuis /ID# 233003, Rotterdam, South Holland
  - Isala /ID# 233031, Zwolle, South Holland
- Poland (4):
  - Szpital Uniwersytecki Nr 1 im. dr Antoniego Jurasza /ID# 232898, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Klinika Pediatrii Gastroenterologii Alergologii i Zywienia Dzieci GUM /ID# 232900, Gdansk, Kuyavian-Pomeranian Voivodeship
  - Poradnia Gastroenterologiczna /ID# 232899, Olsztyn, Kuyavian-Pomeranian Voivodeship
  - Korczowski Bartosz Gabinet Lekarski /ID# 232821, Rzeszow, Kuyavian-Pomeranian Voivodeship
- San Juan Bautista School of Medicine /ID# 232913, Caguas, Puerto Rico
- Instituto Hispalense Pediatria /ID# 232793, Seville, Spain
- Ukraine (4):
  - Kharkiv Regional Childrens Clinical Hospital Gastroent. Centre Kharkiv Natl. Me /ID# 232867, Kharkiv, Cherkasy Oblast
  - Municipal Nonprofit Enterprise Lviv City Children's Clinical Hospital /ID# 232851, Lviv, Cherkasy Oblast
  - Vinnytsya National Medical University Departement of Pediatrics No.1 /ID# 232890, Vinnytsia, Cherkasy Oblast
  - Communal Nonprofit Enterprise City Childrens Clinical Hospital 6 of Dnipro C /ID# 232863, Dnipro
- William Harvey Hospital /ID# 232806, Ashford, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Di Lorenzo C, Khlevner J, Rodriguez-Araujo G, Xie W, Huh SY, Ando M, Hyams JS, Nurko S, Benninga MA, Simon M, Hewson ME, Saps M. Efficacy and safety of linaclotide in treating functional constipation in paediatric patients: a randomised, double-blind, placebo-controlled, multicentre, phase 3 trial. Lancet Gastroenterol Hepatol. 2024 Mar;9(3):238-250. doi: 10.1016/S2468-1253(23)00398-9. Epub 2024 Jan 8. PMID 38211604

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 64 sites, in 7 countries.
Pre-assignment Details: Participants were randomized in a 1:1 ratio for 12 weeks during the double-blind (DB) study intervention period:
  * FC participants received either linaclotide 72 μg or placebo
  * IBS-C participants received either linaclotide 145 μg or 290 μg
  Participants were considered to have completed the study after the DB and Post-Intervention periods. However, the Post-Intervention period was not required for those who enrolled into an open-label, long-term safety study after completing the DB period.
Period: Double-Blind Treatment Period (12 Weeks)
Arm/Group | FC Participants: Placebo | FC Participants: Linaclotide 72 μg | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Started (Randomized) | 164 | 166 | 55 | 53
Randomized and Treated | 164 | 164 | 55 | 53
Completed | 145 | 148 | 52 | 46
Not Completed | 19 | 18 | 3 | 7
Not completed — Lack of Efficacy | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 5 | 1 | 5
Not completed — Lost to Follow-up | 4 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 1 | 0
Not completed — Other, not specified | 4 | 3 | 0 | 1
Not completed — Adverse Event | 2 | 2 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 4 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Post-Intervention Period (1 Week)
Arm/Group | FC Participants: Placebo | FC Participants: Linaclotide 72 μg | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Started | 66 | 75 | 20 | 20
Completed | 65 | 75 | 19 | 20
Not Completed | 1 | 0 | 1 | 0
Not completed — Other, not specified | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | FC Participants: Placebo | FC Participants: Linaclotide 72 μg | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg | Total
Number analyzed (Participants) | 164 | 166 | 55 | 53 | 438
Age, Customized [Count of Participants; unit: Participants]
  6-11 years | 91 | 92 | 22 | 21 | 226
  12-17 years | 73 | 74 | 33 | 32 | 212
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 96 | 31 | 34 | 247
  Male | 78 | 70 | 24 | 19 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 72 | 19 | 17 | 185
  Not Hispanic or Latino | 87 | 94 | 36 | 36 | 253
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 3 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 0 | 0 | 4
  Black or African American | 45 | 42 | 13 | 14 | 114
  White | 114 | 116 | 40 | 35 | 305
  More than one race | 1 | 2 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Functional Constipation (FC) Participants: Change From Baseline in 12-week SBM (Spontaneous Bowel Movement) Frequency Rate (SBMs/Week) During the Study Intervention Period
Description: An SBM is defined as a BM that occurs in the absence of laxative, enema, or suppository use on the calendar day of the bowel movement (BM) or the calendar day before the BM. Assessments of BM characteristics that determine occurrences of SBM (ie, BM frequency and rescue medication use) were measured by using the eDiary completed twice daily (morning and evening) on the eDiary (Electronic Diary) device.
Time Frame: Baseline, up to 12 weeks
Population: Modified Intent-to-Treat Population: all randomized participants who received at least 1 dose of double-blind study intervention. Participants with analysis values at both baseline and postbaseline during the specified time period.
Measure: Least Squares Mean (Standard Error); unit: SBMs
Arm/Group | FC Participants: Placebo | FC Participants: Linaclotide 72 μg
Number analyzed (Participants) | 164 | 164
SBMs | 1.050 (0.187) | 2.220 (0.187)
Statistical Analysis 1: Comparison: FC Participants: Placebo vs FC Participants: Linaclotide 72 μg; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Difference = 1.170, 95% CI 2-sided [0.651 to 1.689], Standard Error of Mean 0.264
Statistical Analysis 2: Comparison: FC Participants: Placebo vs FC Participants: Linaclotide 72 μg; Test type: Superiority; p = 0.4323, ANCOVA — Treatment-by-Age Group Interaction P-value: Interaction P-value base on ANCOVA model with treatment, age group, treatment-by-age group interaction as factors and baseline value as a covariate

2. Primary Outcome: Irritable Bowel Syndrome With Constipation (IBS-C) Participants: 6/12 Weeks APS (Abdominal Pain and SBM) + 2 Responder Rate
Description: 6/12 weeks APS + 2 responder=participant who meets the weekly APS + 2 responder criteria ≥6 of the 12 weeks of the intervention period. Weekly APS +2 responder=participant who has an increase of ≥2 in the SBM weekly rate from baseline, AND a decrease of ≥30% in mean abdominal pain score from baseline, during that study intervention week. Assessments of abdominal pain and BM characteristics that determine occurrences of SBMs were measured by using an eDiary completed twice daily (AM and PM). Assessments of abdominal pain were measured using a 5-point scale where 0=none and 4=a lot. A participant's abdominal pain score=mean of the non-missing abdominal pain scores during the specified period. Responder rate=percentage of participants who were 6/12 weeks APS + 2 responders. A participant had to have ≥4 completed diary days in the analysis week to be considered a responder for that week and was otherwise considered a non-responder for that week.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Number analyzed (Participants) | 53 | 47
percentage of participants | 22.6 | 23.4

3. Secondary Outcome: Functional Constipation (FC) Participants: Change From Baseline in 12-week Stool Consistency During the Study Intervention Period
Description: Stool consistency was measured twice daily, once in the morning and once in the evening eDiary, using the 7-point ordinal pediatric Bristol Stool Form Scale (p-BSFS): Type 1: Looks like small hard lumps or balls, like pebbles; Type 2: Looks like fat sausage shape but lumpy and hard; Type 3: Looks like a sausage but with cracks on it; Type 4: Looks like a sausage or snake, smooth and soft; Type 5: Looks like chicken nuggets, soft smooth blobs; Type 6: Looks like oatmeal, fluffy mushy pieces; Type 7: Looks like a milkshake, watery. A participant's p-BSFS score for the study intervention period was the average of the non-missing p-BSFS scores from the SBMs reported by the participant during the 12-week study intervention period.
Time Frame: Baseline, up to 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FC Participants: Placebo | FC Participants: Linaclotide 72 μg
Number analyzed (Participants) | 132 | 135
units on a scale | 0.685 (0.078) | 1.108 (0.077)
Statistical Analysis 1: Comparison: FC Participants: Placebo vs FC Participants: Linaclotide 72 μg; Test type: Superiority; p = 0.0001, ANCOVA — ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Difference = 0.423, 95% CI 2-sided [0.208 to 0.638], Standard Error of Mean 0.109
Statistical Analysis 2: Comparison: FC Participants: Placebo vs FC Participants: Linaclotide 72 μg; Test type: Superiority; p = 0.4381, ANCOVA — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: Irritable Bowel Syndrome With Constipation (IBS-C) Participants: Change From Baseline in 12-week SBM Frequency Rate (SBMs/Week) During the Study Intervention Period
Description: An SBM is defined as a BM that occurs in the absence of laxative, enema, or suppository use on the calendar day of the BM or the calendar day before the BM. Assessments of BM characteristics that determine occurrences of SBM (ie, BM frequency and rescue medication use) were measured by using the eDiary completed twice daily (morning and evening) on the eDiary (Electronic Diary) device. A participant's SBMs/week for the study intervention period was the average of the non-missing SBMs/week reported by the participant during the 12-week study intervention period.
Time Frame: Baseline, up to 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Number analyzed (Participants) | 53 | 47
SBMs/week | 2.347 (3.3335) | 2.747 (2.8861)

5. Secondary Outcome: Irritable Bowel Syndrome With Constipation (IBS-C) Participants: Change From Baseline in 12-week Abdominal Pain During the Study Intervention Period
Description: Assessments of abdominal pain were measured twice daily, once in the morning and once in the evening eDiary, using a 5-point scale where a score of 0 indicates no abdominal pain scores and a score of 4 indicates a lot of abdominal pain. Assessments of abdominal pain were measured using a 5-point scale where '0' indicates no abdominal pain and '4' indicates a lot of abdominal pain. The participant's abdominal pain score was derived as the mean of the non-missing morning and evening abdominal pain scores during the specified period.
Time Frame: Baseline, up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Number analyzed (Participants) | 53 | 47
units on a scale | -0.837 (0.9313) | -0.837 (0.8809)

6. Secondary Outcome: Irritable Bowel Syndrome With Constipation (IBS-C) Participants: Change From Baseline in 12-week Stool Consistency During the Study Intervention Period
Description: Stool consistency was measured twice daily, once in the morning and once in the evening eDiary, using the 7-point ordinal p-BSFS (pediatric Bristol Stool Form Scale: Type 1: Looks like small hard lumps or balls, like pebbles Type 2: Looks like fat sausage shape but lumpy and hard Type 3: Looks like a sausage but with cracks on it Type 4: Looks like a sausage or snake, smooth and soft Type 5: Looks like chicken nuggets, soft smooth blobs Type 6: Looks like oatmeal, fluffy mushy pieces Type 7: Looks like a milkshake, watery. A participant's p-BSFS score for the study intervention period was the average of the non-missing p-BSFS scores from the SBMs reported by the participant during the 12-week study intervention period.
Time Frame: Baseline, up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Number analyzed (Participants) | 47 | 39
units on a scale | 0.979 (1.2900) | 1.358 (1.1288)

7. Secondary Outcome: Irritable Bowel Syndrome With Constipation (IBS-C) Participants: 6/12 Weeks SBM + 2 Responder Rate
Description: A 6/12 weeks SBM + 2 responder is a participant that meets the weekly SBM + 2 responder criteria for at least 6 out of the 12 weeks of the intervention period. A weekly SBM +2 responder is a participant who has an increase of at least 2 in the SBM weekly rate from baseline, Assessments of BM characteristics that determine occurrences of SBMs (ie, BM frequency and rescue medication use) were measured by using an eDiary completed twice daily (morning and evening). Responder rate is presented as the percentage of participants who were 6/12 weeks SBM + 2 responders.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Number analyzed (Participants) | 53 | 47
percentage of participants | 30.2 | 29.8

8. Secondary Outcome: Irritable Bowel Syndrome With Constipation (IBS-C) Participants: 6/12 Weeks Abdominal Pain Responder
Description: A 6/12 weeks abdominal pain responder is a participant that meets the weekly abdominal pain responder criteria for at least 6 out of the 12 weeks of the intervention period. A weekly abdominal pain responder is a participant who has a decrease of at least 30% in the mean abdominal pain score from baseline, during that study intervention week. Assessments of abdominal pain were measured by using an eDiary completed twice daily (morning and evening) and were measured using a 5-point scale where '0' indicates no abdominal pain and '4' indicates a lot of abdominal pain. The participant's abdominal pain score was derived as the mean of the non-missing abdominal pain scores during the specified period. Responder rate is presented as the percentage of participants who were 6/12 weeks abdominal pain responders.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
Number analyzed (Participants) | 53 | 47
percentage of participants | 49.1 | 42.6

ADVERSE EVENTS:
Time Frame: Up to 13 weeks
Description: All randomized participants
Arm/Group | FC Participants: Linaclotide 72 μg | FC Participants: Placebo | IBS-C Participants: Linaclotide 145 μg | IBS-C Participants: Linaclotide 290 μg
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/164 | 0/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 2/166 | 2/164 | 0/55 | 0/53
Other Adverse Events (participants affected / at risk) | 11/166 | 10/164 | 7/55 | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FC Participants: Linaclotide 72 μg (N=166) | FC Participants: Placebo (N=164) | IBS-C Participants: Linaclotide 145 μg (N=55) | IBS-C Participants: Linaclotide 290 μg (N=53)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FAECALOMA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FC Participants: Linaclotide 72 μg (N=166) | FC Participants: Placebo (N=164) | IBS-C Participants: Linaclotide 145 μg (N=55) | IBS-C Participants: Linaclotide 290 μg (N=53)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 6 (6) | 3 (3) | 4 (4) | 4 (4)
COVID-19 (Infections and infestations) | 4 (4) | 5 (5) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT04026113/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT04026113/SAP_001.pdf